CLINICAL TRIAL: NCT01207830
Title: A Single Center Feasibility Trial of the Safety and Efficacy of the ValenTx Endo Bypass System in Obese Subjects
Brief Title: Feasibility Trial of ValenTx Endo Bypass System of the ValenTx Endo Bypass System in Obese Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ValenTx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LA 2.2
Record Dates: First submitted 2010-09-21; First posted 2010-09-23 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Obesity
Keywords: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endo Bypass (Experimental): Subjects implanted with the investigational ValenTx Endo Bypass System
  Interventions: Device: Endo Bypass System

INTERVENTIONS:
Device: Endo Bypass System — Subject is implanted with the device for up to 3 years.
  Other Names: Valentx; EBS

SUMMARY:
The purpose of this study is to provide initial clinical data to support the feasibility of use of the ValenTx Endo Bypass system in enhancing weight loss and co-morbidity resolution in morbidly obese subjects

DETAILED DESCRIPTION:
This is a single center, open label, feasibility study whose major aim is to determine the feasibility (based on safety, efficacy and device performance) of the ValenTx Endo Bypass system with the replaceable sleeve. Also, the use of a tag replacement device may be developed and implemented should individual attachment tags need replaced following the initial implant.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 55 years of age
* Subject has a BMI >35 kg/m2 and <= 50 kg/m2, with or without co-morbid conditions(s)
* Documented failure with non-surgical weight loss methods
* Willing to comply with study procedures and visit schedule
* Willing and able to provide informed consent

Exclusion Criteria:

* Pregnancy or intention of becoming pregnant within the study duration (Women of childbearing potential participating in the study must have a negative serum pregnancy test result at screening and use a medically acceptable form of contraception. Medically acceptable forms of contraception include oral contraceptives, injectable or implantable methods, intrauterine devices, or properly used double-barrier contraception, eg condom plus diaphragm. If screening pregnancy test is done greater than 7 days before implant, women of childbearing potential must have another serum pregnancy test result before implantation. Any woman becoming pregnant during the treatment period must withdraw from the study)
* Endoscopic lesions such as important hiatal hernia, gastric or duodenal ulcer, atresias or stenosis, polyps of the stomach
* Subject with potential upper gastrointestinal bleeding such as esophageal or gastric varices, Mallory-Weis syndrome or congenital or acquired intestinal telangiectasia
* Past history of esophageal or gastric/GI surgery, obstruction, adhesive peritonitis, or large hiatal hernia (> 3 cm)
* IBS, unexplained intermittent vomiting, severe abdominal pain or chronic constipation within 60 days of study day 0
* Unexplained anaemia, Pancreatitis, Portal hypertension, Esophagitis or Barrett's esophagus, known gallstones or anomalies of the GI tract
* Any bodily infections within 30 days of study day 0 (implant day)
* Prolonged steroid use
* Hep C or HIV positive
* Known allergies to any of the device materials
* Use of weight loss medication within 2 months prior to enrollment and throughout the study period
* Recent or ongoing cancer, history of severe renal, hepatic, cardiovascular or pulmonary disease or transplants
* Inability to tolerate anti-inflammatory medications
* Evidence of psychiatric problems or dietary habits that would contraindicate study treatment
* Active drug or alcohol addiction within 12 months of enrollment and throughout the study duration
* Prior history of inflammatory diseases of the GI tract, (e.g., esophagitis, varices, gastric or duodenal ulceration, or Crohn's disease; congenital or acquired GI anomalies, e.g., bowel strictures)
* Ongoing treatment with anticoagulants, steroids, aspirin, NSAIDs, or other gastric irritants within 1 month prior to enrollment and throughout the study period
* Participation in previous (within 60 days of study day 0) or ongoing clinical trial or current or past usage (within 60 days of study day 0) of investigation drug or other device

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-03; Primary Completion 2011-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Device-related adverse events | 1-3 years

SECONDARY OUTCOMES:
Device Performance | 1-3 years

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Rumbaut, M.D., Principal Investigator — Hospital San Jose Tec
Locations (1):
- Hospital San Jose Tec de Monterrey, Monterrey, Mexico

REFERENCES:
- [Derived] Sandler BJ, Rumbaut R, Swain CP, Torres G, Morales L, Gonzales L, Schultz S, Talamini MA, Jacobsen GR, Horgan S. One-year human experience with a novel endoluminal, endoscopic gastric bypass sleeve for morbid obesity. Surg Endosc. 2015 Nov;29(11):3298-303. doi: 10.1007/s00464-015-4081-5. Epub 2015 Jan 29. PMID 25631114